CLINICAL TRIAL: NCT07179471
Title: "Fake Carbs" Practice in the Glycemic Outcomes in Children and Adolescents Using AID System: A Cross-over Observational Study
Brief Title: Fake Carbs Practice With AID System - MiniMed 780G in Children and Adolescents With T1D.
Acronym: CHeatAID
Status: Recruiting | Type: Observational
Sponsor: Maria Chatzipsalti (Other)
Responsible Party: Sponsor-Investigator, Maria Chatzipsalti, Pediatrician and Pediatric Endocrinologist-Diabetologist, Athens General Children's Hospital "Pan. & Aglaia Kyriakou"
Organization: Athens General Children's Hospital "Pan. & Aglaia Kyriakou" (Other)
Other Study IDs: 10862
Record Dates: First submitted 2025-07-03; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: AID System; MiniMed 780G; Fake carbs; AHCL System
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (FC1): 20 individuals who use 'fake carbohydrates' to correct hyperglycemia will continue using this strategy for two weeks.
- Group 2 (FC2):: 20 individuals who use 'fake carbohydrates' to correct hyperglycemia will discontinue this strategy for two weeks

SUMMARY:
Hybrid Closed Loop (HCL) systems, such as the MiniMed 780G, have significantly improved glycemic outcomes in Type 1 Diabetes (T1D) management. The MiniMed 780G, an Advanced Hybrid Closed Loop (AHCL) system, features autocorrection boluses and unique insulin adjustment technologies. While effective, the system requires user input for meal announcements. Some individuals attempt to "trick" the system by entering "fake carbs" to prompt additional insulin corrections. However, clinical evidence suggests this practice does not improve glycemic outcomes.

This study, conducted in Athens, Greece, will involve 40 children and adolescents (ages 7-18) with Type 1 Diabetes who have been using the MiniMed 780G system for over 6 months. The open-label, crossover design explores the impact of 'fake carbohydrates' on glycemic control. Participants will be split into two groups: one starts with 'fake carbohydrates' and then stops, while the other does the reverse. Over two weeks, their glycemic outcomes will be monitored and compared, with exclusions for severe diabetes complications or serious diabetic events

This study hypothesizes that using "fake carbs" does not enhance glycemic control. Findings are expected to provide evidence-based insights to optimize diabetes management and improve clinical guidance for HCL system users.

DETAILED DESCRIPTION:
Aim of the Study To compare glycemic control outcomes in individuals with T1D using the MiniMed™ 780G system during periods when 'fake carbohydrates' are used versus periods when this strategy is not employed.

Definition: Fake Carbohydrates As a Fake Carbs practice is defined the practice when the user enters fake quantity of carbohydrates in order to trigger the system to suggest and deliver a bolus insulin with the aim to correct hyperglycemia.

Study Design and Participants This is a prospective, open-label, randomized, crossover trial conducted at the Diabetes Center of the General Hospital "P. & A. Kyriakou" in Athens, Greece.

Sample Size

* Total Participants: 40 children and adolescents
* Age Range: 7-18 years Inclusion Criteria
* Diagnosis of T1D
* Using the MiniMed™ 780G system for ≥6 months
* Habitual use of fake carbohydrates in daily management Exclusion Criteria
* Severe diabetes-related complications
* Recent episodes of diabetic ketoacidosis (DKA) or severe hypoglycemia Randomization and Group Allocation

Participants will be randomized into two groups based on their prior use of fake carbohydrates:

Group 1 (FC1): Continue using fake carbohydrates for 2 weeks, followed by discontinuation for 2 weeks.

Group 2 (FC2): Discontinue use of fake carbohydrates for 2 weeks, followed by resumption for 2 weeks.

Each intervention phase will be preceded by a 2-week run-in period to allow algorithm adaptation. A 2-week washout period between crossover phases will follow the same adaptation rationale.

Baseline and Ongoing Assessments

* Clinical and Demographic Data
* Age, sex, T1D duration, weight, height
* HbA1c measured via HPLC (Menarini) on a single analyzer All data retrieved from hospital electronic medical records

MiniMed™ 780G System Data

Review of pump settings during run-in phase

Settings optimized using:

* Target glucose: 100 mg/dL
* Active Insulin Time: 2 hours

Fake Carbohydrates Logbook

Participants will maintain a log recording:

* Time, amount, and context of fake carbohydrate entries
* Real meals and blood glucose levels
* Any episodes of hypoglycemia following fake CHO entries

Outcome Measures

* Primary Outcome Time in Range (TIR 70-180 mg/dL) over each 2-week intervention phase
* Secondary Outcomes Time below range (<70 mg/dL) and time above range (>180 mg/dL) Total daily insulin dose Frequency and severity of hypoglycemia System usage data (auto-mode %, correction boluses) Number and frequency of meal and fake CHO entries Adverse events (e.g., severe hypoglycemia, DKA)

Data Collection Tools CareLink™ Software: Used for glycemic data at baseline, week 2, and week 4 Participant logbooks for qualitative assessment of FC practices

Data Analysis Within-subject comparisons will be conducted due to crossover design Descriptive statistics for demographic and baseline characteristics Paired t-tests or Wilcoxon signed-rank tests for primary and secondary outcomes Repeated-measures ANOVA for longitudinal outcomes

Expected Impact This study will provide the first structured evaluation of the widely used but clinically unverified practice of entering 'fake carbohydrates' in AHCL systems. It will inform clinicians on whether this strategy improves or undermines glycemic control and support evidence-based recommendations for pump users and healthcare providers.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 7-18 years
* T1D >6 months
* on MiniMed 780G system in automode.

Exclusion Criteria:

* Participants with significant diabetes complications
* Participants with severe episode of diabetic ketoacidosis in the last 6 months
* Participants with hypoglycemia in the last 6 months.

Ages: 7 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — All
Study Population: Participants (Age 7-18 years) with T1D using MiniMed 780G system for 6 months at least.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Time In Range | 2 weeks
  Change between groups in blood glucose in Time in Range -TIR ( defined as 70-180 mg/dl) (%)
Change in Time in Tight Range | 2 weeks
  Change between groups in time in blood glucose in Tight Range -TITR ( defined as 70-140 mg/dl) (%)
Change in Time Below Range | 2 weeks
  Change between groups in blood glucose in Time Below Range- TBR (defined as <54mg/dl) (%)

SECONDARY OUTCOMES:
Changes between groups in GMI | 2 weeks
  Changes between groups in Glucose Management Indicator (GMI, %).
Changes in Time Above Range | 2 weeks
  Changes between groups in blood glucose in Time Above Range (%)
Change in mean sensor glucose | 2 weeks
  Change between groups in mean sensor glucose (SG, mg/dl).
Change in Standard Deviation of glucose | 2 weeks
  Changes between groups in Standard Deviation of glucose (SD, mg/dl)
Changes in Coefficient of Variation for glucose | 2 weeks
  Changes between groups in Coefficient of Variation for glucose (CV, %)
Changes in number of announced carbs | 2 weeks
  Changes between groups in number of announced carbs (gr/day)
Changes in total daily insulin dose | 2 weeks
  Changes between groups in total daily insulin dose (TDD, units/day).
Changes in insulin Auto-basal rate | 2 weeks
  Changes between groups in insulin Auto-basal rate (%)
Changes in insulin Auto-correction | 2 weeks
  Changes between groups in insulin Auto-correction rate (%)
Changes in insulin Manual bolus | 2 weeks
  Changes between groups in insulin Manual bolus (%)
Changes in number of severe hypoglycemia episodes | 2 weeks
  Changes between groups in number of severe hypoglycemia episodes, defined as as the ones requiring medical assistance.
Changes in the number of diabetic ketoacidosis (DKA) events | 2 weeks
  Changes between the groups in the number of diabetic ketoacidosis (DKA) events , defined as:
  * Blood glucose >200 mg/dl
  * Venous pH <7.3 or serum bicarbonate <15 mmol/L
  * Ketonemia (β-hydroxybutyrate ≥3 mmol/L) (β-hydroxybutyrate ≥3 mmol/L)

CONTACTS AND LOCATIONS:
Locations (3):
- Greece (3):
  - Athens General Children's Hospital "Pan. & Aglaia Kyriakou", Athens, Attica
  - Athens, Attiki, Athens, Attica
  - Diabetes Center, Athens, Attica

IPD SHARING:
Plan to Share IPD: Undecided
Willing to share upon request.